CLINICAL TRIAL: NCT07066917
Title: Mechanisms of Response and Resistance to Innovative Treatments in Patients With Locally Advanced or Metastatic Breast Cancer
Acronym: PANDORA
Status: Recruiting | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HE_11PDR/24
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Breast Cancer
Keywords: mBC; biomarkers; ADCs; immunotherapy; PARPi; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Peripheral blood will be collected for ctDNA analysis and germline mutation testing before initiation of treatment and at disease progression. FFPE tissue and H&E slided will be collected for whole exome sequencing and digital pathology respectively at diagnosis and at disease progression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ADCs: Patients receiving treatment with an Antibody-Drug conjugate (e.g Trastuzumab-Deruxtecan, Sacituzumab-Govitecan)
- ICIs: Patients receiving treatment with an immune checkpoint inhibitor (ICI) (e.g pembrolizumab)
- PARPi: Patients receiving treatment with a PARP inhibitor (e.g Olaparib)

SUMMARY:
Ample evidence has highlighted the significant clinical benefit of novel therapies for many patients with advanced breast cancer (aBC). The use of CDK inhibitors, antibody-drug conjugates (ADCs), immune checkpoint inhibitors (ICIs), and PARP inhibitors as first-line or subsequent treatments has improved progression-free survival (PFS) rates compared to conventional therapies. In selected cases, these treatments have also increased overall survival (OS), reshaping the therapeutic landscape for advanced breast cancer.

However, several key questions remain unanswered. For example, what should be the first-line treatment when multiple effective options are available? Determining the optimal sequence of drugs in successive lines of therapy is another major challenge. Furthermore, the development of resistance to treatment and the occurrence of severe adverse events that may lead to early discontinuation or fatal outcomes are pressing concerns.

That said, identifying robust predictive biomarkers of response or resistance is crucial for ensuring that patients receive the most effective treatment while avoiding unnecessary exposure to therapies that could cause harm without benefit. Additionally, when multiple effective options exist, selecting the optimal treatment algorithm for each patient based on clinical, pathological, and molecular biomarkers is essential.

We herein, aim at employing high throughput methodologies, such as Whole Exome Sequencing, circulating tumour DNA (ctDNA) analysis, digital pathology and radiomics analyses, as well as real-world data obtained both from patients records for the training of a ML-based algorithm that can predict response or resistance to a specific treatment, based on the genetic make-up of the patient and the molecular profile of the tumour.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be 18 years of age and older
* Histologically confirmed, advanced breast cancer.
* Diagnosis of i) hormone receptor positive and/or ii) HER2-positive or -low or iii) triple negative breast cancer (TNBC).
* Patients will be included in the analysis after receiving at least one treatment cycle.

Exclusion Criteria:

* Diagnosis of early breast cancer at time of enrollment
* Unwillingness to provide informed consent
* Unwillingness to provide biological specimen
* Lack of comprehensive clinical data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with histologically confirmed, advanced breast cancer of one of the following subtypes: i) Hormone receptor positive and/or ii) HER2-positive or -low or iii) triple negative breast cancer (TNBC)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Through study completion, 5 years
  Correlation of genetic and molecular/circulating biomarkers with PFS, with PFS defined as the time from enrollment to disease progression or death
Overall Survival (OS) | Through study completion, 5 years
  Correlation of genetic and molecular/circulating biomarkers with OS, with OS defined as the time from date of metastatic diagnosis to last follow-up (36 months, post enrollment) or death
Objective Response Rate (ORR) | Through study completion, 5 years
  Correlation of genetic and molecular biomarkers with response to treatment

SECONDARY OUTCOMES:
Evaluation of AI-predictive algorithm | Through study completion, 5 years
  Evaluation of the efficiency of the AI-predictive algorithm, by determining key metrics such as sensitivity and specificity

CONTACTS AND LOCATIONS:
Overall Officials: Elena Fountzilas, MD, PhD, Principal Investigator — Hellenic Cooperative Oncology Group
Locations (5):
- Greece (5):
  - University General Hospital "ATTIKON", 2nd propedeutic dept. of Internal Medicine, Athens
  - "MITERA" Hospital, Dept. of Medical Oncology, Athens
  - Metropolitan Hospital, 2nd Dept. of Medical Oncology, Athens
  - Metropolitan Hospital, 4th Dept. of Medical Oncology, Athens
  - St. Luke's Hospital, Dept. of Medical Oncology, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartzberg L, Kim ES, Liu D, Schrag D. Precision Oncology: Who, How, What, When, and When Not? Am Soc Clin Oncol Educ Book. 2017;37:160-169. doi: 10.1200/EDBK_174176. PMID 28561651
- [Background] D'Arienzo A, Verrazzo A, Pagliuca M, Napolitano F, Parola S, Viggiani M, Caputo R, Puglisi F, Giuliano M, Del Mastro L, Arpino G, De Laurentiis M, Montemurro F. Toxicity profile of antibody-drug conjugates in breast cancer: practical considerations. EClinicalMedicine. 2023 Jul 27;62:102113. doi: 10.1016/j.eclinm.2023.102113. eCollection 2023 Aug. PMID 37554126
- [Background] Guidi L, Pellizzari G, Tarantino P, Valenza C, Curigliano G. Resistance to Antibody-Drug Conjugates Targeting HER2 in Breast Cancer: Molecular Landscape and Future Challenges. Cancers (Basel). 2023 Feb 10;15(4):1130. doi: 10.3390/cancers15041130. PMID 36831473
- [Background] Fenton MA, Tarantino P, Graff SL. Sequencing Antibody Drug Conjugates in Breast Cancer: Exploring Future Roles. Curr Oncol. 2023 Nov 29;30(12):10211-10223. doi: 10.3390/curroncol30120743. PMID 38132377
- [Background] Litton JK, Rugo HS, Ettl J, Hurvitz SA, Goncalves A, Lee KH, Fehrenbacher L, Yerushalmi R, Mina LA, Martin M, Roche H, Im YH, Quek RGW, Markova D, Tudor IC, Hannah AL, Eiermann W, Blum JL. Talazoparib in Patients with Advanced Breast Cancer and a Germline BRCA Mutation. N Engl J Med. 2018 Aug 23;379(8):753-763. doi: 10.1056/NEJMoa1802905. Epub 2018 Aug 15. PMID 30110579
- [Background] Robson M, Im SA, Senkus E, Xu B, Domchek SM, Masuda N, Delaloge S, Li W, Tung N, Armstrong A, Wu W, Goessl C, Runswick S, Conte P. Olaparib for Metastatic Breast Cancer in Patients with a Germline BRCA Mutation. N Engl J Med. 2017 Aug 10;377(6):523-533. doi: 10.1056/NEJMoa1706450. Epub 2017 Jun 4. PMID 28578601
- [Background] Schmid P, Adams S, Rugo HS, Schneeweiss A, Barrios CH, Iwata H, Dieras V, Hegg R, Im SA, Shaw Wright G, Henschel V, Molinero L, Chui SY, Funke R, Husain A, Winer EP, Loi S, Emens LA; IMpassion130 Trial Investigators. Atezolizumab and Nab-Paclitaxel in Advanced Triple-Negative Breast Cancer. N Engl J Med. 2018 Nov 29;379(22):2108-2121. doi: 10.1056/NEJMoa1809615. Epub 2018 Oct 20. PMID 30345906
- [Background] Cortes J, Rugo HS, Cescon DW, Im SA, Yusof MM, Gallardo C, Lipatov O, Barrios CH, Perez-Garcia J, Iwata H, Masuda N, Torregroza Otero M, Gokmen E, Loi S, Guo Z, Zhou X, Karantza V, Pan W, Schmid P; KEYNOTE-355 Investigators. Pembrolizumab plus Chemotherapy in Advanced Triple-Negative Breast Cancer. N Engl J Med. 2022 Jul 21;387(3):217-226. doi: 10.1056/NEJMoa2202809. PMID 35857659
- [Background] Bardia A, Hurvitz SA, Tolaney SM, Loirat D, Punie K, Oliveira M, Brufsky A, Sardesai SD, Kalinsky K, Zelnak AB, Weaver R, Traina T, Dalenc F, Aftimos P, Lynce F, Diab S, Cortes J, O'Shaughnessy J, Dieras V, Ferrario C, Schmid P, Carey LA, Gianni L, Piccart MJ, Loibl S, Goldenberg DM, Hong Q, Olivo MS, Itri LM, Rugo HS; ASCENT Clinical Trial Investigators. Sacituzumab Govitecan in Metastatic Triple-Negative Breast Cancer. N Engl J Med. 2021 Apr 22;384(16):1529-1541. doi: 10.1056/NEJMoa2028485. PMID 33882206
- [Background] Rugo HS, Bardia A, Marme F, Cortes J, Schmid P, Loirat D, Tredan O, Ciruelos E, Dalenc F, Gomez Pardo P, Jhaveri KL, Delaney R, Valdez T, Wang H, Motwani M, Yoon OK, Verret W, Tolaney SM. Overall survival with sacituzumab govitecan in hormone receptor-positive and human epidermal growth factor receptor 2-negative metastatic breast cancer (TROPiCS-02): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2023 Oct 21;402(10411):1423-1433. doi: 10.1016/S0140-6736(23)01245-X. Epub 2023 Aug 23. PMID 37633306
- [Background] Modi S, Saura C, Yamashita T, Park YH, Kim SB, Tamura K, Andre F, Iwata H, Ito Y, Tsurutani J, Sohn J, Denduluri N, Perrin C, Aogi K, Tokunaga E, Im SA, Lee KS, Hurvitz SA, Cortes J, Lee C, Chen S, Zhang L, Shahidi J, Yver A, Krop I; DESTINY-Breast01 Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Positive Breast Cancer. N Engl J Med. 2020 Feb 13;382(7):610-621. doi: 10.1056/NEJMoa1914510. Epub 2019 Dec 11. PMID 31825192
- [Background] Modi S, Jacot W, Yamashita T, Sohn J, Vidal M, Tokunaga E, Tsurutani J, Ueno NT, Prat A, Chae YS, Lee KS, Niikura N, Park YH, Xu B, Wang X, Gil-Gil M, Li W, Pierga JY, Im SA, Moore HCF, Rugo HS, Yerushalmi R, Zagouri F, Gombos A, Kim SB, Liu Q, Luo T, Saura C, Schmid P, Sun T, Gambhire D, Yung L, Wang Y, Singh J, Vitazka P, Meinhardt G, Harbeck N, Cameron DA; DESTINY-Breast04 Trial Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Low Advanced Breast Cancer. N Engl J Med. 2022 Jul 7;387(1):9-20. doi: 10.1056/NEJMoa2203690. Epub 2022 Jun 5. PMID 35665782